CLINICAL TRIAL: NCT03178565
Title: The Effects of Mechanical Insufflation-exsufflation for Airway Mucus Clearance Among Mechanically Ventilated ICU Patients: a Randomized Trial
Brief Title: The Effects of Mechanical Insufflation-exsufflation on Airway Mucus Clearance in the ICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Moinhos de Vento (Other)
Responsible Party: Principal Investigator, Augusto Savi, PhD, Hospital Moinhos de Vento
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CoughAssist trial
Record Dates: First submitted 2017-04-21; First posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Respiratory Failure
Keywords: Respiratory Failure; Mechanical Ventilation; Mechanical insufflation-exsufflation; Airway mucus clearance
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Mechanically ventilated patients will be randomized to receive respiratory physiotherapy using a mechanical insufflation-exsufflation device (intervention group) or to receive standard respiratory physiotherapy without the use of a mechanical insufflation-exsufflation device (control group).
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Respiratory physiotherapy using a mechanical insufflation-exsufflation device (CoughAssist)
  Interventions: Other: Mechanical insufflation-exsufflation
- Control Group (Active Comparator): Respiratory physiotherapy according standard of care - without the use of a mechanical insufflation-exsufflation device.
  Interventions: Other: Standard Respiratory Physiotherapy

INTERVENTIONS:
Other: Mechanical insufflation-exsufflation — The mechanical insufflation-exsufflation device will be connected in the orotracheal tube. Four series of insufflation-exsufflation will be conducted. Each serie will be composed by 10 cycles of alternated insufflation (40 cmH2O) and exsufflation (- 40 cmH2O).
  Other Names: CoughAssist
  Arms: Intervention Group
Other: Standard Respiratory Physiotherapy — Standard chest physiotherapy will be conducted through bilateral thoracic maneuvers (percussion and vibration) followed by manual hyperinflation using a manual resuscitator bag.
  Arms: Control Group

SUMMARY:
The present study aims to evaluate the effect of mechanical insufflation-exsufflation on airway mucus clearance among mechanically ventilated ICU patients. A parallel group randomized clinical trial will be conducted in a single mixed medical-surgical ICU of a tertiary hospital in Southern Brazil. Adult ICU patients with a length of mechanical ventilation >24 hours will be evaluated for eligibility. Patients will be randomized in a 1:1 ratio to receive respiratory physiotherapy using a mechanical insufflation-exsufflation device (intervention group) or standard respiratory physiotherapy without the use of the mechanical insufflation-exsufflation device (control group). The primary outcome is the amount of aspirated respiratory mucus (weight in grams) 5 minutes after the finish of respiratory physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Admission to the ICU
* Length of mechanical ventilation > 24 hours
* Stable ventilatory and hemodynamic status defined by positive end- expiratory pressure ≤ 8 cm H2O, inspiratory oxygen fraction ≤ 40%, ratio of arterial oxygen partial pressure to fractional inspired oxygen ≥ 150, respiratory rate ≤ 35 breaths per minute, heart rate ≤ 130 beats per minute and systolic blood pressure between 90 and 160 mmHg.

Exclusion Criteria:

* Patients with primary neuromuscular disease.
* Patients in exclusive paliative care.
* Patients with contraindications to the use of mechanical insufflation- Exsufflation device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Amount of aspirated secretion | This outcome will be verified 5 minutes after the completion of the study intervention on the day of subject enrollment.
  Single measure of weight in grams of the aspirated secretion 5 minutes after the study intervention (mechanical insufflation-exsufflation or standard respiratory physiotherapy).

SECONDARY OUTCOMES:
Static lung compliance | This outcome will be verified 5 minutes after the completion of the study intervention on the day of subject enrollment.
  Single measure of the static lung compliance in mL/cm H2O
Airway resistance | This outcome will be verified 5 minutes after the completion of the study intervention on the day of subject enrollment.
  Single measure of the airway resistance in cm H2O/L/s

CONTACTS AND LOCATIONS:
Overall Officials: Marcio Camillis, Principal Investigator — Hospital Moinhos de Vento
Locations (1):
- Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferreira de Camillis ML, Savi A, Goulart Rosa R, Figueiredo M, Wickert R, Borges LGA, Galant L, Teixeira C. Effects of Mechanical Insufflation-Exsufflation on Airway Mucus Clearance Among Mechanically Ventilated ICU Subjects. Respir Care. 2018 Dec;63(12):1471-1477. doi: 10.4187/respcare.06253. Epub 2018 Jul 17. PMID 30018175